CLINICAL TRIAL: NCT04061746
Title: Cellular Therapy for Type 1 Diabetes Using Mesenchymal Stem Cells
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Hongjun Wang, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00085542; R01DK118529-01A1 (NIH)
Record Dates: First submitted 2019-08-16; First posted 2019-08-20 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: mesenchymal stem cells; diabetes; autoantibodies; C-peptide; Type 1 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Plasmalyte A; Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A Treatment (Experimental): 2.5 x 10^6 MSC per kg will be infused intravenously on Day 1
  Interventions: Biological: Mesenchymal Stem Cells (MSCs)
- Group B Placebo (Placebo Comparator): Plasmalyte with 0.5% Human Serum Albumin will be infused intravenously on Day 1
  Interventions: Other: Placebo Infusion (Plasmalyte A with 0.5% human serum albumin)

INTERVENTIONS:
Biological: Mesenchymal Stem Cells (MSCs) — Patients in Group A will receive a single MSCs infusion
  Arms: Group A Treatment
Other: Placebo Infusion (Plasmalyte A with 0.5% human serum albumin) — Patients in Group B will receive a single infusion of placebo (Plasmalyte A with 0.5% human serum albumin)
  Arms: Group B Placebo

SUMMARY:
The goal of this study is to determine the safety and efficacy of fresh metabolically active allogeneic umbilical cord-derived mesenchymal stromal cells (UC-MSCs) for the treatment of new-onset type 1 diabetes (T1D) and to understand the mechanisms of protection. If proven effective, such a strategy can be used as a therapeutic option for T1D patients and potentially other autoimmune disorders.

DETAILED DESCRIPTION:
This study seeks to find and enroll participants between the ages of 18 to 40 with new onset Type 1 diabetes (T1D) within 6 months of the first dose of insulin. T1D is an autoimmune disease in which T cells attack and destroy insulin-secreting pancreatic β cells leading to insulin deficiency and hyperglycemia in patients. Life-long insulin therapy is the major treatment option. However, insulin therapy is not a cure and a safer and more effective therapy is needed.

Mesenchymal Stromal Cells (MSCs) have emerged as a novel biopharmaceutical approach for many disorders. MSCs are a cellular product that can be derived from a patient's own body (autologous) or from a donor (allogeneic). This study will obtain MSCs from umbilical cords at the time of delivery from normal women who have been extensively screened for infectious diseases. These cells produced at the MUSC Center for Cellular therapy will be used within 3 passages after collection.

Evidence from animal models and clinical trials suggests that MSC infusion suppresses autoimmune and inflammatory diseases such as T1D. One clear message from these trials is that MSCs are effective at suppressing autoimmunity and seem generally safe. This study will measure safety and efficacy of MSCs over the course of 1 year.

ELIGIBILITY:
Inclusion criteria:

* A new diagnosis of T1D based on the ADA criteria within 6 months of randomization.
* Male and female between the ages of 18 and 40
* Mentally stable and able to comply with the procedures of the study protocol
* Positivity for at least one T1D-associated autoantibody, such as GAD, IA-2 or ZnT8 autoantibodies
* At screening, patients must have residual β cell function with a stimulated peak C-peptide >0.2 nmol/l during a 2 hour MMTT
* Must be willing to comply with "intensive diabetes management" (* See diabetes management at MUSC below) as directed by the participant's clinician with the goal of maintaining blood glucose as close to normal as possible
* Subject must be willing to comply with the schedule of study visits and protocol requirements
* Subject with normal laboratory values of: White blood cell counts: between 4,500 to 11,000 per microliter; Platelet counts: 140,000 to 450,000 platelets per microliter of blood; Serum creatinine range is 0.6-1.3 mg/dL, Hepatic function: ALT 5 to 55 units per liter (U/L), AST 5 to 48 U/L.

Exclusion criteria:

* Evidence of retinopathy at baseline based on ophthalmologic examination or medical record review.
* Body Mass Index < 14 or >35
* Presence of malignancy
* Subject has abnormally high lipid levels that exceeds > 3 times the upper limit of normal for LDL cholesterol or triglycerides
* Subject has blood pressure greater than 160 mmHg systolic or 100 mmHg diastolic at time of consent
* Subject is being treated for severe active infection of any type
* A female subject who is breast-feeding, pregnant, or intends to become pregnant during the study.
* Subject with clinically relevant uncontrolled medical condition not associated with diabetes (e.g. severe psychiatric, hematologic, renal, hepatic, neurologic, cardiac, or respiratory disorder)
* Subjects with HgbA1c >12%, and/or fasting blood glucose >270 mg/dL and/or frequent episodes of hypoglycemia (>2 episodes per week of blood glucose levels <60 mg/dL).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-02-27 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
12 month Change in C-peptide area under the curve after a 2-hour MMTT | 1 year (plus or minus 30 days) after infusion
  Change in beta cell function

SECONDARY OUTCOMES:
6 Month Change in C-Peptide area under the curve after a 2-hour MMTT | 6 months (plus or minus 14 days) after infusion
  Change in beta cell function
6 Month peak C-peptide after a 2-hour MMTT | 6 months (plus or minus 14 days) after infusion
  Change in beta cell function
1 year peak C-peptide after a 2-hour MMTT | 1 year (plus or minus 30 days) after infusion
  Change in beta cell function
Change in 24-hour insulin dose per kilogram between baseline and 1 year measurements | 1 year (plus or minus 30 days) after infusion
  Change in beta cell function

OTHER OUTCOMES:
Fasting and postprandial blood glucose levels after MSC infusion | 0 - 72 Hours
  Change in beta cell function
Changes in basal C-peptide and hemoglobin A1c | Over the course of 1 year (0, 1, 3, 6, 12 months)
  Change in beta cell function
Change in serum glucagon levels | Over the course of 1 year (0, 1, 3, 6, 12 months)
  Change in alpha cell function
Insulin secretion rate | Over the course of 1 year (0, 1, 3, 6, 12 months)
  Change in beta cell function
Changes in islet autoanitbodies | Over the course of 1 year (0, 1, 3, 6, 12 months)
  Change in autoantibody presence or titer
Change in beta cell death measurements | Over the course of 1 year (0, 1, 3, 6, 12 months)
  Determination of the mechanism of action
Change in blood T-reg number and function | Over the course of 1 year (0, 1, 3, 6, 12 months)
  Determination of the mechanism of action
Change in autoantigen specific T-cell response | Over the course of 1 year (0, 1, 3, 6, 12 months)
  Determination of the mechanism of action
Change in blood autoreactive B cell number, B cell survival, and function | Over the course of 1 year (0, 1, 3, 6, 12 months)
  Determination of the mechanism of action
Changes in mRNA expression in peripheral blood mononuclear cells after treatment | Over the course of 1 year (0, 1, 3, 6, 12 months)
  Determination of the mechanism of action
Changes in serum cytokine levels after treatment | Over the course of 1 year (0, 1, 3, 6, 12 months)
  Determination of the mechanism of action

CONTACTS AND LOCATIONS:
Overall Officials: Hongjun Wang, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No